CLINICAL TRIAL: NCT05749913
Title: Cognitive Load of Activity Participation Scale (CLAP): Development and Validation
Status: Terminated | Type: Observational
Why Stopped: The research has been transferred to another project leader.
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202301132RIND
Record Dates: First submitted 2023-02-20; First posted 2023-03-01 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2024-05

CONDITIONS: Aging
Keywords: participation; cognitive activities; cognitive load

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 14 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Normal: 1. Participants living in the community.
  2. No vision or hearing impairment.
  3. No severe depression, or other neurological/mental disorders affecting cognitive function.
- Subjective Cognitive Decline, SCD: 1. The Montreal Cognitive Assessment (MoCA) score >22
  2. Use two questions to screen: "Compared with the previous situation, do you have memory problems?", "Has your family or relatives ever thought that you have memory problems compared with the previous situation?", the answer to both questions is yes.
  3. Geriatric Depression Scale-Short Form (GDS-S) score <8
- Mild Cognitive Impairment, MCI: 1. MCI diagnosed by neurologists or psychiatrists: the diagnosis of MCI is mainly in accordance with the revised consensus version of the diagnostic criteria (Winblad et al., 2004), that is, memory function score is 1.5 standard deviations below the value for age- and education-related norms on the third edition of Wechsler Memory Scale.
  2. MoCA: with a range of scores of 17-23(>17 , <23) (Trzepacz et al., 2015)
  3. Geriatric Depression Scale-Short Form (GDS-S) score <8
- Mild Dementia: 1. has met the criteria of dementia
  2. at the early stages

SUMMARY:
In this study, we develop and validate the " Cognitive Load of Activity Participation Scale" (CLAPs) to measure the frequency and the perceived levels of cognitive load of the elderly participating in various cognitive activities and as a reference for intervention and behavioral Indicators for lifestyle modifications to preventing and delaying dementia.

DETAILED DESCRIPTION:
The purpose of this study in the first year is to develop the first version of the CLAPs by literature review, focus group discussion, expert validity, etc., to collect the typical participation in daily and housework activities, social leisure and entertainment, work and learning activities of the elderly. And we also evaluate the level of cognitive load of subjective feelings when individuals participate in activities. In the second year, the aim is to complete the final version of the CLAPs, which is expected to collect 300 subjects in the first version. According to the results, we analyze and select the items and verify the psychometric characteristics, including test-retest reliability and construct validity (factor analysis and convergent validity). In the third year, we will recruit 150 people over 65 with different cognitive levels, including subjective cognitive decline, mild cognitive impairment, and mild dementia, to validate the discriminant validity. The CLAPs will provide an understanding of the cognitive activity profile of the person and as a guide for interventions and an outcome measure.

ELIGIBILITY:
Inclusion Criteria:

* Years 1 and 2 of study:

  1. Participants living in the community, aged 65 or above.
  2. No vision or hearing impairment, able to communicate and read in Mandarin and Taiwanese.
  3. No severe depression, or other neurological/mental disorders affecting cognitive function.
* Third year of study:

Subjective Cognitive Degeneration (SCD):

1. Participants living in the community, aged 65 or above.
2. No vision or hearing impairment, able to communicate and read in Mandarin and Taiwanese.
3. The Montreal Cognitive Assessment (MoCA) score >22
4. Use two questions to screen: "Compared with the previous situation, do you have memory problems?", "Has your family or relatives ever thought that you have memory problems compared with the previous situation?", the answer to both questions is yes.
5. Geriatric Depression Scale-Short Form (GDS-S) score <8

Mild Cognitive Impairment (MCI):

1. Participants living in the community, aged 65 or above.
2. No vision or hearing impairment, able to communicate and read in Mandarin and Taiwanese.
3. MCI diagnosed by neurologists or psychiatrists: the diagnosis of MCI is mainly in accordance with the revised consensus version of the diagnostic criteria (Winblad et al., 2004), that is, memory function score is 1.5 standard deviations below the value for age- and education-related norms on the third edition of Wechsler Memory Scale.
4. MoCA: with a range of scores of 17-23(>17, <23) (Trzepacz et al., 2015)
5. Geriatric Depression Scale-Short Form (GDS-S) score <8

Mild Dementia:

1. Participants living in the community, aged 65 or above.
2. No vision or hearing impairment, able to communicate and read in Mandarin and Taiwanese.
3. Those who have met the diagnostic criteria for mild dementia are referred by the neurologist or psychiatrist.

Exclusion Criteria:

* Years 1 and 2 of study:

  1. Have a history of diseases related to cognitive degeneration (for example: acute stroke, brain injury, unconsciousness, etc.), and those diagnosed with organic nerve damage, brain function disorders, and related neurology.
  2. People with serious mental illness or behavior problems.
* Third year of study:

SCD:

1. Cognitive changes caused by other mental, neurological diseases, or substance abuse, etc.
2. Has met the diagnostic criteria of MCI or dementia
3. Those who are unable to complete the cognitive test due to visual, auditory, physical or cognitive impairment

MCI:

1. Cognitive changes caused by other mental, neurological diseases, or substance abuse, etc.
2. Has met the diagnostic criteria for dementia.
3. Those who are unable to complete the cognitive test due to visual, auditory impairment

Mild Dementia:

1. Cognitive changes caused by other mental, neurological diseases, or substance abuse, etc.
2. Those who cannot accept the cognitive test because they are visually or hearing impaired, or have serious physical disease and behavioral problems.

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Normal: No vision or hearing impairment, and no severe depression, or other neurological/mental disorders affecting cognitive function
  SCD: Use two questions to screen: "Compared with the previous situation, do you have memory problems?", "Has your family or relatives ever thought that you have memory problems compared with the previous situation?", the answer to both questions is yes.
  MCI: meet the criteria of Mild Cognitive Impairment
  Mild Dementia: meet the criteria of dementia
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2023-03-16 (Actual); Primary Completion 2023-05-25 (Actual); Study Completion 2023-05-25 (Actual)

PRIMARY OUTCOMES:
The Montreal Cognitive Assessment(MoCA) | 10-15 mins
  The Montreal Cognitive Assessment (MoCA) is a sensitive tool for screening cognitive function in the early stages of cognitive degeneration.
Geriatric Depression Scale-Short Form (GDS-S) | 5-7 minutes
  There are 15 questions for elderly in GDS-S used for screening depression state. It takes 5-7 minutes to complete.

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Fen Mao, M.S., Principal Investigator — National Taiwan University Hospital
Locations (1):
- College of Medicine, National Taiwan University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
ethical issue